CLINICAL TRIAL: NCT00565071
Title: Parasite-based Diagnosis for Malaria in Uganda: Feasibility and Cost-Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Department for International Development, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Institute of Public Health, Prof. Fred Nuwaha, MD, PhD, Makerere University School of Public Health, Makerere University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/HD20/4758U
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Fever; Malaria
Keywords: Cost-effectiveness; Diagnosis; Treatment; Malaria
MeSH Terms: conditions — Fever; Malaria; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Field microscopy (Other): Field microscopy is the main method of malaria diagnosis
  Interventions: Device: Field microscopy and Paracheck Pf®
- Paracheck Pf® device (Other): Paracheck Pf® device (Rapid Diagnostic Test) is the main method for malaria diagnosis
  Interventions: Device: Field microscopy and Paracheck Pf®
- Presumptive diagnostic method (No Intervention)

INTERVENTIONS:
Device: Field microscopy and Paracheck Pf® — Malaria diagnosis based on microscopy and or Paracheck Pf®. Artemether/Lumefantrine (20mg/120mg) is first-line drug in all arms
  Arms: Field microscopy; Paracheck Pf® device

SUMMARY:
The purpose of this study is to compare the cost-effectiveness of treating malaria based on three methods of diagnosis (rapid test, microscopy and presumptive diagnosis) among patients attending level three government health centres located in areas of low and high transmission intensities in Uganda. The study hypotheses are: in both low and high transmission areas, cost-effectiveness of malaria treatment with Artemether-Lumefantrine will be improved by the adoption of rapid diagnostic tests when compared with presumptive diagnosis or microscopy; and the difference between the cost-effectiveness of Artemether-Lumefantrine treatment following rapid diagnostic test or microscopy versus presumptive diagnosis will be greatest in low transmission areas.

DETAILED DESCRIPTION:
The development of drug resistance in malaria parasites lead the Uganda Ministry of Health (MoH) to change the first-line anti-malarial treatment from the cheap Chloroquine/Sulfadoxine-Pyrimethamine combination to a more expensive Artemether-Lumefantrine. The MoH recommends treatment of all fever cases as malaria within 24 hours of illness with first-line drug. Under this policy, patients who do not have malaria but present with febrile illness will receive Coartem® resulting in significant drug wastage. With the increased cost of first-line drugs, this wastage places a substantial and potentially remediable burden on the health budget. As such, there is a need to gauge whether more accurate malaria diagnosis through microscopy and/or rapid diagnostic tests, might improve the cost-effectiveness of the new treatment regimes.

Specific objectives

1. To assess the feasibility of rapid test and microscopy in diagnosis of malaria at health centre III.
2. To compare the cost-effectiveness of treating malaria with Artemether- Lumefantrine based on microscopy, rapid test and presumptive diagnosis in different transmission intensities
3. To assess whether introduction of malaria parasite-based diagnosis (rapid test or microscopy) at government Health Centre III improves the overall cost-effectiveness of outpatient management of febrile illness

Sample size determination The sample size was determined using standard formula. Estimating the sensitivity of either test to be 90%, Zα =1.96 and after stratifying for age (<5 years and ≥5 years), the calculated sample is 272 per health centre. Therefore, the total number of patients for 6 health centres in two districts = 6 x 272 = 1632.

Baseline: Baseline data was collected on the current malaria treatment practices; clinicians' view of malaria diagnosis; concerns towards the new treatment; and health centre staffing. Geographical locations of all visited government health centres was recorded using Germin etrex global positioning system (Germin International Inc., Olathe, USA). At six selected health centres, social and demographic data was collected from 613 patients.

Implementation of intervention: The main intervention is comprised of three malaria diagnostic approaches: presumptive diagnosis, field microscopy and rapid test (Paracheck Pf® device - Orchid Biomedical Systems, Goa, India). Each of these approaches was randomly allocated to a health centre. The first-line drug used is Artemether/Lumefantrine (20mg/120mg) (Novartis, Switzerland).

Consenting subjects are consecutively enrolled at the point when the attending clinician suspects that they have uncomplicated malaria. Where microscopy is the main diagnostic method, thick and thin blood smears are prepared per patient enrolled. Where rapid test is the main method, all patients are tested. One hundred patients per health centre are randomly selected to provide blood specimens for validation using expert microscopy and PCR as "gold standard." After enrolment, patients are systematically tracked until departure from the health centre. Patients are followed up on the seventh day of treatment to assess their clinical improvement. Those who fail to return on the scheduled date are traced from their homes on the eighth day.

Follow-up activities include: documentation of drugs prescribed and or dispensed; clinically assess the patient's status in comparison to Day 0; perform further tests including PCR if the patient does not show improvement; pill counting of drugs remaining - if the patient has not completed the dose; documentation of reasons for not completing dose; and documentation if the patient bought the prescribed drugs that were out of stock on Day 0.

Effectiveness is measured as the number of patients commencing treatment with Artemether/Lumefantrine. However, patients are followed up and effectiveness also measured on the 7th day of treatment indicated by their clinical improvement. The feasibility of the diagnostic methods is ongoing from the March 2010 to date.

ELIGIBILITY:
Inclusion Criteria:

* Suspected uncomplicated malaria infection
* Consent to participate

Exclusion Criteria:

* Pregnancy (policy recommends quinine for treatment of malaria in pregnancy)

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102087 (Estimated)
Dates: Start 2006-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic test validity; unit cost per malaria case diagnosed and treated with Artemether-Lumefantrine; total savings associated with treatment of confirmed malaria cases; compliance with directives for use of rapid test or microscopy | 18 months

SECONDARY OUTCOMES:
unit cost of non-malaria febrile treatment; therapeutic behaviour in light of pressure to prescribe antimalarials | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Fred Nuwaha, MD, PhD, Study Chair — Department of Disease Control and Environmental Health, Makerere Universtiy School of Public Health
Locations (1):
- Bushenyi and Iganga districts - Government Health Cetres level III, Bushenyi and Iganga, Uganda

REFERENCES:
- [Derived] Batwala V, Magnussen P, Nuwaha F. Challenges to implementation of artemisinin combination therapy policy in Uganda. Int Health. 2010 Dec;2(4):262-8. doi: 10.1016/j.inhe.2010.07.002. PMID 24037867
- [Derived] Batwala V, Magnussen P, Mirembe J, Mulogo E, Nuwaha F. Timing of malaria messages for target audience on radio airwaves. Malar J. 2012 Aug 20;11:283. doi: 10.1186/1475-2875-11-283. PMID 22905781
- [Derived] Batwala V, Magnussen P, Nuwaha F. Antibiotic use among patients with febrile illness in a low malaria endemicity setting in Uganda. Malar J. 2011 Dec 20;10:377. doi: 10.1186/1475-2875-10-377. PMID 22183039
- [Derived] Batwala V, Magnussen P, Nuwaha F. Comparative feasibility of implementing rapid diagnostic test and microscopy for parasitological diagnosis of malaria in Uganda. Malar J. 2011 Dec 19;10:373. doi: 10.1186/1475-2875-10-373. PMID 22182758
- [Derived] Batwala V, Magnussen P, Hansen KS, Nuwaha F. Cost-effectiveness of malaria microscopy and rapid diagnostic tests versus presumptive diagnosis: implications for malaria control in Uganda. Malar J. 2011 Dec 19;10:372. doi: 10.1186/1475-2875-10-372. PMID 22182735
- [Derived] Batwala V, Magnussen P, Nuwaha F. Are rapid diagnostic tests more accurate in diagnosis of plasmodium falciparum malaria compared to microscopy at rural health centres? Malar J. 2010 Dec 2;9:349. doi: 10.1186/1475-2875-9-349. PMID 21126328